CLINICAL TRIAL: NCT04368884
Title: A Prospective, Longitudinal, Observational Study to Assess the Seroconversion Status of Front Line Health Care Workers and Comparison With the Suspected or Confirmed Cases of COVID-19 Patients at Max Health Care (Project D)
Brief Title: Assess the Seroconversion Status of Health Care Workers Suspected or Confirmed Cases of COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: Covid-19/MHC-2/2020
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Covid-19
Keywords: Seroconversion; Healthcare Workers; COVID-19
MeSH Terms: conditions — COVID-19; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples are being stored at -70C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthcare workers: The healthcare workers who are being tested for COVID-19 would be included in this group
- OPD patients: Individuals outside from the hospital who are coming for the COVID-19 testing will be included in this group
- IPD COVID-19 cases: Admitted positive cases of COVID-19 in the hospital will be included in this group

SUMMARY:
A large number of Health Care Workers (HCWs) would be potentially getting exposed to COVID19. Some of them would be asymptomatic or may get subclinical symptoms. Our HCW would have higher exposure and possibly higher seroconversion either symptomatic or with clinical symptoms than the general population. This study is aimed to understand the rate of seroconversion states at different stages of exposure. It is crucial to collect baseline immune status and the early immunological changes that might occur in asymptomatic or symptomatic health care workers and to compare that with the suspected or confirmed cases by following them for six weeks.

DETAILED DESCRIPTION:
This prospective observational, longitudinal study is being conducted at Max Super Specialty Hospital, Saket, New Delhi. Below mentioned are the study objectives-

Primary Objectives

* To determine the extent of infection in the healthcare workers (HCW) of a tertiary care hospital in India, by determining the seropositivity
* To compare immune changes that might occur in healthcare workers who are asymptomatic or symptomatic with the proven positive cases in OPD or IPD at Max hospital.

Secondary Objectives

* To determine the fraction of asymptomatic or subclinical infections
* To understand the seroconversion status at different stages of exposure to front line HCW

The study population would include all employees of Max Hospitals, Delhi-NCR, who have been tested for COVID-19. Samples and data of the COVID positive patients admitted in the hospital will also be collected and OPD patients coming to the hospital for COVID-19 testing will be one of the study subsets.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers of Max Hospital, irrespective of age and gender OR
* COVID-19 positive patients admitted in the hospital OR
* Out-patients getting tested for COVID-19

Exclusion Criteria:

* Refusal to give informed consent, or contraindication to venipuncture.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All employees of Max Hospital, Saket and Smart, New Delhi, who are coming to the hospital, working in the COVID ward or the nearby wards, and who would agree to participate will be recruited in this study including those who are being tested in suspicion of COVID-19. Samples and data of the COVID positive patients admitted in the hospital will also be collected. OPD patients coming to the hospital for COVID-19 testing will be one of the study subsets.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Development of antibodies | 4-8 weeks
  Samples will be assessed for the presence of IgG and IgM

CONTACTS AND LOCATIONS:
Overall Officials: Sujeet Jha, MRCP (U.K), Principal Investigator — Max Healthcare Institute Ltd.
Locations (1):
- Max Super Speciality Hospital, A Unit of Devki Devi Foundation, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet prepared an IPD sharing protocol at this stage. Data might be shared if requested.